CLINICAL TRIAL: NCT04110548
Title: Emotion and Craving Regulation Among Individuals With Internet Gaming Disorder: Cognitive Appraisal and Mindfulness Capacities
Brief Title: Emotion and Craving Regulation Among Individuals With Internet Gaming Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, bnuzhounan, Associated Professor, Beijing Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ER&CR_IGD
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Internet Gaming Disorder; Emotion Regulation
Keywords: Emotion and craving regulation
MeSH Terms: conditions — Internet Addiction Disorder; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HCs on Emotion Regulation (Experimental): Participants are screened using the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5), Young's online Internet addiction test (YIAT), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), and so on. They are instructed to complete the emotion regulation task on the computer.
  Interventions: Procedure: Emotion Regulation Task
- IGDs on Emotion Regulation (Experimental): Participants are screened using the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5), Young's online Internet addiction test (YIAT), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), and so on.They are instructed to complete the emotion regulation task on the computer.
  Interventions: Procedure: Emotion Regulation Task
- IGDs on Craving Regulation (Experimental): Participants are screened using the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5), Young's online Internet addiction test (YIAT), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), and so on. They are instructed to complete the craving regulation task on the computer.
  Interventions: Procedure: Craving Regulation Task

INTERVENTIONS:
Procedure: Emotion Regulation Task — Participants are instructed to complete the emotion assessment after Look or Decrease the neutral or negative pictures. The "Decrease" asks the participants to use "cognitive reappraisal" or "mindfulness" strategies to decrease the intensity of emotion, whereas the "Look" asks the participants to look naturally at the picture. First, the "look" or "decrease" is displayed on the computer for 2 s. Then, a neutral or negative picture is presented on the screen for 7s. Finally, participants will rate the intensity of their emotion for 4s. Then, they have 1s-3s to relax before the next trial. In the meantime, Skin conductance activities will be recorded using a constant voltage with 1-cm 3 AgAg/Cl electrodes attached to the medial phalanx surfaces of the middle and index fingers of the nondominant hand.
  Arms: HCs on Emotion Regulation; IGDs on Emotion Regulation
Procedure: Craving Regulation Task — Participants are instructed to complete the craving assessment after Look or Decrease the neutral or gaming pictures. The "Decrease" asks the participants to use "cognitive reappraisal" or "mindfulness" strategies to decrease the intensity of craving, whereas the "Look" asks the participants to look naturally at the picture. First, the "look" or "decrease" is displayed on the computer for 2 s. Second, a neutral or gaming picture is presented on the screen for 7s. Third, participants rate the intensity of their craving for 4s. Then, they have 1s-3s to relax before the next trial. In the meantime, Skin conductance activities will be recorded using a constant voltage with 1-cm 3 AgAg/Cl electrodes attached to the medial phalanx surfaces of the middle and index fingers of the nondominant hand.
  Arms: IGDs on Craving Regulation

SUMMARY:
To investigate the potential deficits in emotion and craving regulation capacities of drug-naïve young adults with Internet gaming disorder as compared with healthy controls.

DETAILED DESCRIPTION:
The purpose of this study is to examine the differences in young adults' capacities of utilizing cognitive appraisal versus mindfulness to regulate negative emotions and/or craving in response to negative affective stimuli or gaming cues, respectively. This project will be conducted in Beijing, China.

ELIGIBILITY:
Inclusion Criteria:

Internet gaming disorders (IGD):

1, DSM-5 recommended diagnosis of Internet gaming disorder :

1. the scores of the 9 items of DSM-5 recommended diagnosis for Internet gaming disorder ≥ 5.
2. engagement in popular Internet games (e.g. Arena of Valor, League of Legends and Player Unknown's Battle Grounds) for over 20 hours per week for a minimum of 12 months.

2, the scores of the Y-IAT(Young-Internet addiction Test) ≥ 50

Healthy controls (HCs): DSM-5 scores less than 5 and less than 20 hours gaming time per week.

Exclusion Criteria:

current or history of use of illegal substances and gambling; current or history of psychiatric or neurological illness; current use of psychotropic medications; being left-handed.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Behavioral outcome | 30- 40 minutes after training
  Participants' ratings of negative emotion and their skin conductance levels (SCL).
Behavioral outcome | 40- 60 minutes after training
  Participants' ratings of negative emotion and their skin conductance levels (SCL).
Behavioral outcome | 60- 80 minutes after training
  Participants' ratings of cravings and their skin conductance levels (SCL).

CONTACTS AND LOCATIONS:
Overall Officials: Nan Zhou, PhD, Principal Investigator — Beijing Normal University
Locations (1):
- Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yip SW, Gross JJ, Chawla M, Ma SS, Shi XH, Liu L, Yao YW, Zhu L, Worhunsky PD, Zhang J. Is Neural Processing of Negative Stimuli Altered in Addiction Independent of Drug Effects? Findings From Drug-Naive Youth with Internet Gaming Disorder. Neuropsychopharmacology. 2018 May;43(6):1364-1372. doi: 10.1038/npp.2017.283. Epub 2017 Nov 20. PMID 29154365
- [Background] Westbrook C, Creswell JD, Tabibnia G, Julson E, Kober H, Tindle HA. Mindful attention reduces neural and self-reported cue-induced craving in smokers. Soc Cogn Affect Neurosci. 2013 Jan;8(1):73-84. doi: 10.1093/scan/nsr076. Epub 2011 Nov 22. PMID 22114078